CLINICAL TRIAL: NCT02710903
Title: IL29 and IL28B Variants Associated With Periodontal Disease Pathogenesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-0637; 5K23DE025093-02 (NIH); 5K23DE025093-03 (NIH)
Record Dates: First submitted 2015-12-08; First posted 2016-03-17 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Periodontitis
Keywords: Periodontitis; SNP; Pathogenesis; IL29; IL28B
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy with Dominant IL28B and IL29 (Experimental): Stent-induced biofilm overgrowth model will be used in dominant IL28B and IL29 allelic with probing depths (PD) ≤4mm, no evidence of inter proximal clinical attachment loss (CAL), and <20% of sites with bleeding on probing (BOP).
  Interventions: Procedure: Stent-induced biofilm overgrowth
- Periodontal Disease with Dominant IL28B and IL29 (Experimental): Stent-induced biofilm overgrowth model will be used in dominant IL28B and IL29 allelic with the presence of at least four periodontal sites with PD ≥ 5mm, evidence of interproximal CAL, and ≥20% of sites with BOP.
  Interventions: Procedure: Stent-induced biofilm overgrowth
- Healthy with IL28B and/or IL29 SNP variants (Experimental): Stent-induced biofilm overgrowth model will be used in IL28B or IL29 SNP variants with PD ≤4mm, no evidence of interproximal CAL, and <20% of sites with BOP.
  Interventions: Procedure: Stent-induced biofilm overgrowth
- Periodontal Disease with IL28B and/or IL29 SNP variants (Experimental): Stent-induced biofilm overgrowth model will be used in IL28B or IL29 SNP variants with the presence of at least four periodontal sites with PD ≥ 5mm, evidence of interproximal CAL, and ≥20% of sites with BOP.
  Interventions: Procedure: Stent-induced biofilm overgrowth

INTERVENTIONS:
Procedure: Stent-induced biofilm overgrowth — Customized stents will be fabricated for each subject. Stents will be fabricated to resemble an acrylic mouth-guard but extended to cover approximately 2mm over gingival margins. Stents will form a seal and rest on the gingiva, but will be relieved on the tooth and tissue side except for the occlusal surfaces to avoid disturbing plaque or gingival tissues. Acrylic stents will abstained from brushing and flossing teeth in one maxillary and one mandibular posterior sextant during a three- week period. Patients will be monitored for safety every week and after the induction of experimental biofilm overgrowth through 21 days

SUMMARY:
A maximum of 220 subjects with a minimum of 25 years will be recruited and examined for this 1-7 visit, up to 35 days research study: Subjects will be genotyped to identify variants of the interleukin-29 (IL29) and interleukin-28B (IL28B) genes and placed in one of the 4 groups: 50 subjects with dominant allelic variants with healthy periodontium, 50 subjects with dominant allelic variants with periodontitis, 50 subjects with IL29 (rs30461) or any of IL28B (rs11083519; rs8105790; rs8099917) single nucleotide polymorphism's (SNP) variants and healthy periodontium, and 50 subjects with IL29 (rs30461) or any of IL28B (rs11083519; rs8105790; rs8099917) SNP variants and periodontitis. Visits will consist of outpatient procedures including oral examinations, oral prophylaxis or periodontal scaling and root planing, collection of gingival crevicular fluid, dental plaque, saliva, and blood samples. Analysis will include salivary DNA isolation and pyrosequencing to determine IL29 and IL28B genotype, mediator analysis of gingival crevicular fluid, dendritic cell differentiation and inflammatory mediator analysis, and whole-genome shotgun sequencing plaque analysis. Clinical outcomes will include measurements of periodontal disease progression and inflammation, such as clinical attachment level (CAL), pocket depth (PD), bleeding on probing (BOP), gingival index (GI), and plaque index (PI).

Primary Objective: To determine the impact of IL29 and IL28B SNP variants on periodontal disease expression and local inflammatory response during stent-induced biofilm overgrowth.

Secondary Objective: To evaluate in vitro the impact of IL29 and IL28B SNP variants on cell-mediated, innate inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have read, understood and signed an informed consent form in English.
* Subjects must be able and willing to follow study procedures and instructions in English.
* Subjects must be non-Hispanic Caucasian.
* Subjects must be adult males or females with a minimum of 25 years (inclusive).
* Subjects must present with at least 20 teeth in the functional dentition, excluding third molars.
* Subjects must have at least 3 teeth in each posterior sextant.
* Subjects must be in good general health.
* Subjects must present with one of the following four categories to be considered for enrollment:
* Dominant IL28B and IL29 allelic with PD ≤4mm, no evidence of interproximal CAL, and <20% of sites with BOP.
* Dominant IL28B and IL29 allelic with the presence of at least four periodontal sites with PD ≥ 5mm, evidence of interproximal CAL, and ≥20% of sites with BOP.
* IL28B or IL29 SNP variants with PD ≤4mm, no evidence of interproximal CAL, and <20% of sites with BOP.
* IL28B or IL29 SNP variants with the presence of at least four periodontal sites with PD ≥ 5mm, evidence of interproximal CAL, and ≥20% of sites with BOP

Exclusion Criteria:

* Chronic disease with oral manifestations including diabetes mellitus.
* Current smoker or one that has stopped smoking less than 2 years prior to enrollment.
* Gross oral pathology other than the periodontal disease.
* Treatment with antibiotics for any medical or dental condition within 1 month prior to the screening examination.
* Chronic treatment (i.e., two weeks or more) with any medication known to affect periodontal status (e.g., phenytoin, calcium antagonists, cyclosporin, coumadin, non-steroidal anti-inflammatory drugs, aspirin) within one month of the screening examination.
* Ongoing medications initiated less than three months prior to enrollment (i.e., medications for chronic medical conditions must be initiated at least three months prior to enrollment).
* Significant organ disease including impaired renal function, heart murmur, history of rheumatic fever or valvular disease, or any bleeding disorder.
* Infectious diseases such as hepatitis, HIV or tuberculosis.
* Anemia or other blood dyscrasias.
* Anticoagulant therapy or drugs, such as heparin or warfarin.
* Severe unrestored caries, or any condition that is likely to require antibiotic treatment over the trial.
* Pregnant, or expect to become pregnant within the next several months.
* Females of child-bearing capacity must be willing to have pregnancy test to confirm they are not pregnant.
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-05; Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Change in pocket depth (mm) | 21 days
Change in clinical attachment level (mm) | 21 days
Change in plaque index (0-3) | 21 days
Change in bleeding on probing (Yes/No) | 21 days
Change in gingival crevicular fluid interleukin-1 beta (GCF IL-1b) | 21 days
Change in gingival crevicular fluid prostaglandin E2 (GCF PGE2) | 21 days
Change in gingival crevicular fluid interleukin-29 (GCF IL-29) | 21 days
Change in gingival crevicular fluid interleukin-28B (GCF IL-28B) | 21 days
Change in gingival index (0-4) | 21 days
Composition of the microbiota oral flora | 21 days
Change in gingival crevicular fluid interleukin-6 (GCF IL-6) | 21 days

SECONDARY OUTCOMES:
Change in interleukin-29 expression in dendritic cells at day 35 | 35 days
Change in interleukin-28B expression in dendritic cells at day 35 | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Jim Beck, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States